CLINICAL TRIAL: NCT03617991
Title: Functional and Self-reported Outcomes in Participants With a History of Musculoskeletal
Brief Title: Functional and Self-reported Outcomes in Participants With a History of Musculoskeletal Knee Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johanna M. Hoch (Other)
Responsible Party: Sponsor-Investigator, Johanna M. Hoch, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB #43308
Record Dates: First submitted 2018-07-06; First posted 2018-08-07 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Anterior Cruciate Ligament Injury; Anterior Cruciate Ligament Rupture
Keywords: rehabilitation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Participants will be provided an 8-week home exercise program that they will complete. The participants will also be provided all of the equipment. An investigator will contact them weekly to ensure compliance and send You Tube videos with new Phases.
  Interventions: Other: Exercise Group
- Control Group (No Intervention): The control group will be contacted weekly to check on health status.

INTERVENTIONS:
Other: Exercise Group — An 8-week home exercise program will be given to the participants. The program is designed to have four phases, progressed every two weeks. The participants will receive and email from study personnel every two weeks with new videos detailing the progression of exercises. The participants will be given all of the equipment to complete the exercises. The exercises will include balance and strength training exercises for the core and lower extremity.
  Arms: Exercise Group

SUMMARY:
Negative outcomes impact individuals with a history of ACL reconstruction (ACLR) despite completion of formal rehabilitation and clearance to return to physical activity (PA). Focused exercises and targeted health education may improve these negative outcomes and increase quality of life. The purpose of this study is determine the effects of an 8-week rehabilitation program on strength, sensorimotor function, functional performance and patient-reported outcomes in patients with a history of ACLR. A secondary aim will be to identify baseline PA levels and dietary intake patterns in these individuals. Participants will complete standard knee radiographs and all baseline measures, and resume normal activities of daily living for one-week while wearing an accelerometer to quantify PA levels and complete two, 24-hour dietary recalls to examine dietary patterns. After one-week, participants will come back to the laboratory and complete the pre-intervention assessments prior to randomization to the exercise or control group. After 8-weeks, participants will complete all outcome assessments 24-48 hours, 1-month and 3-months post exercise completion. The investigators hypothesize the intervention group will have significantly better outcomes post-intervention compared to the control group. In addition, the investigators hypothesize areas of educational and behavioral intervention related to PA engagement and dietary strategies to support weight management will be needed.

ELIGIBILITY:
Inclusion Criteria:

* History of unilateral ACL reconstruction,
* History of injuring their knee playing or training for sports (recreational or organized),
* Have been cleared to participate in activity, do not have radiographic evidence of post-traumatic osteoarthritis,
* Are free of neurological disorders, cardiopulmonary disease or any other condition that may impact their ability to participate

Exclusion Criteria:

* ACL reconstruction >10 years,
* Injury to either lower extremity within the last 6-weeks,
* Surgery to either limb within the last year,
* A BMI > 30

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Joint Specific Self-Reported Function | Baseline, pre-intervention (one week later just prior to the initiation of the intervention), 24-48 hours post-intervention, 1-month and 3-months post
  Participants will complete the Knee Injury and Osteoarthritis Outcome (KOOS) survey to assess self-reported knee joint function across five domains (pain, symptoms, activities of daily living, sport and recreation, and quality of life). The questionnaire will include 42 questions across the domains, that are scored on a 5-point Likert scale. Each subscale is scored separately, and range from 0-100 (100=perfect self-reported knee function). The scores are transformed for each subscale as follows: 100-(actual raw score x 100)/ possible raw score. Participants will complete the survey at the time of consent, one week later just prior to the initiation of the intervention, up to 48 hours after completion of the intervention, then at 1 and 3 month follow up visits. Data will be presented longitudinally as the change in self-reported function over the duration of the study, up to three months.

SECONDARY OUTCOMES:
Change in Fear Avoidance Behaviors | Baseline, pre-intervention (one week later just prior to the initiation of the intervention), 24-48 hours post-intervention, 1-month and 3-months post
  Participants will complete the Fear Avoidance Belief Questionnaire (FABQ) to evaluate fear avoidance during activities of sport and physical activity. The FABQ is a 15-item survey, scored on a 6-point Likert scale where 6 is completely agree and 0 is completely disagree. There are 5 items in the FABQ-PA section and 10-items in the Sport section. Higher scores indicate elevate levels of fear avoidance beliefs. Participants will complete the survey at time of consent, one week later just prior to the initiation of the intervention, up to 48 hours after completion of the intervention, then at 1 and 3 month follow up visits. Data will be presented longitudinally as the change of fear avoidance beliefs over the duration of the study and up to three months after the intervention.
Change in General Health-Related Quality of Life | Baseline, pre-intervention (one week later just prior to the initiation of the intervention), 24-48 hours post-intervention, 1-month and 3-months post
  Participants will complete the modified Disablement in the Physically Active Scale (mDPA) to evaluate general health related quality of life. This questionnaire will include 16 questions across two domains (physical and mental) and is scored on a 5-point Likert scale, where 0 indicates no problem and 4 indicates severe problem. The mDPA-physical component has 12-items, and scores can range from 0-48 while there are 4 items on the mDPA-mental and scores range from 0-16. Higher scores indicate decreased health-related quality of life. Scores are simply added for each component to get a final score. Participants will complete the survey at the time of consent, one week later just prior to the initiation of the intervention, up to 48 hours after completion of the exercise regimen (intervention), then at 1 and 3 month follow up visits. Data will be presented longitudinally as the change in self-reported health related quality of life over the duration of the study, up to three months.
Change in Knee related Self-Efficacy | Baseline, pre-intervention (one week later just prior to the initiation of the intervention), 24-48 hours post-intervention, 1-month and 3-months post
  Participants will complete the Knee Self-Efficacy Scale (KSES) to evaluate their knee-related self-efficacy. This questionnaire will include 22 questions, each scored on a 0-10 scale where 0-not at all certain and 10-very certain. There are four sections: Daily activities, sport and leisure activities, physical activities and knee function in the future. The sum of the items is calculated and then divided by the total number of items to get a total score. Higher scores indicate greater levels of knee self-efficacy. Participants will complete the survey at the time of consent, one week later just prior to the initiation of the intervention, up to 48 hours after completion of the exercise regimen (intervention), then at 1 and 3 month follow up visits. Data will be presented longitudinally as the change in knee-related self-efficacy through the duration of the study, up to three months.
Change in Fear of Movement | Baseline, pre-intervention (one week later just prior to the initiation of the intervention), 24-48 hours post-exercise completion, 1-month post, 3-months post
  Participants will complete the Tampa Scale of Kinesiophobia-11(TSK-11) to evaluate their fear of movement/re-injury. This is an 11-item scale scored on a 4-point Likert scale where 1=strongly disagree and 4= strongly agree. The total score is a sum of all items, with scores ranging from 11-44. Participants will complete the survey at the time of consent, one week later just prior to the initiation of the intervention, up to 48 hours after completion of the intervention, then at 1 and 3 month follow up visits. Data will be presented longitudinally as the change in fear of movement and re-injury over the duration of the study, up to three months.
Change in Dynamic Balance | Baseline, pre-intervention (one week later just prior to the initiation of the intervention), 24-48 hours post-intervention, 1-month and 3-months post
  Participants will complete the Y-balance test as a measure of dynamic balance. This assessment will require the participant to stand on a plastic box, and push a plastic box as far as they can in three different directions. This will be done on both feet, and a measure of dynamic balance will be determined for all three directions. Participants will complete this measure at time of consent, one week later just prior to the initiation of the intervention, up to 48 hours after completion of the intervention, then at 1 and 3 month follow up visits. Data will be presented longitudinally as the change in dynamic balance over the duration of the study, up to three months.
Change in Static Balance | Baseline, pre-intervention (one week later just prior to the initiation of the intervention), 24-48 hours post-intervention, 1-month and 3-months post
  Participants will complete the Balance Error Scoring System to evaluate their static balance. This will include the participants standing barefoot, on one limb, with their eyes closed while an investigator counts their errors. The participants will complete this assessment at the time of consent, one week later just prior to the initiation of the intervention, up to 48 hours after completion of the intervention, and then at 1 and 3 month follow-up visits. Data will be presented longitudinally as the change in static balance over the duration of the study, up to three months.
Change in Functional Abilities | Baseline, pre-intervention )(one week later just prior to the initiation of the intervention), 24-48 hours post-intervention, 1-month and 3-months post
  Participants will complete 4 functional hops (4 hop series) to evaluate their functional abilities. The functional hop series will include the: triple hop for distance where the patient will be asked to hop three times, on one leg, as far as they can; the single-leg hop for distance where the participant will be asked to hop as far as they can on one leg; the crossover hop for distance where the patient will be asked to hop back and forth for a certain distance and the six-meter timed hop where the patient will be asked to hop as fast as they can for six meters. Participants will complete these tests at the time of consent, one week later just prior to the intervention, up to 48 hours after completion of the intervention, then at 1 and 3 month follow-up visits. Data will be presented longitudinally as the change in function over the duration of the study, up to three months.
Change in Landing Errors | Baseline, pre-intervention (one week later just prior to the initiation of the intervention), 24-48 hours post-intervention, 1-month and 3-months post
  Participants will complete the Landing Error Scoring System to evaluate their landing errors. This will involve standing on a 30cm box, and jumping out and up four times. The investigator will assess the number of errors at each jump. Participants will complete this assessment at the time of consent, one week later just prior to initiation of the intervention, up to 48 hours after completion of the intervention, then at 1 and 3 month follow-up visits. Data will be presented longitudinally as the change in landing errors over the duration of the study and up to 3 months.
Change in Strength | Baseline, pre-intervention (one week later just prior to the initiation of the intervention), 24-48 hours post-intervention, 1-month and 3-months post
  Participants will have their knee and hip muscle strength tested using a hand held device. The measurements of strength will include: knee extension, knee flexion, hip abduction, hip adduction, hip flexion and hip extension. Participants will complete these measurements at the time of consent, one week later just prior to the initiation of the intervention, 48-hours after completion of the intervention, then at 1 and 3 month follow-up visits. Data will be presented longitudinally as the change in strength measurements over the duration of the study, up to three months.

CONTACTS AND LOCATIONS:
Overall Officials: Johanna M Hoch, PhD, ATC, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No